CLINICAL TRIAL: NCT06137534
Title: The Effect of Proprioceptive Neuromuscular Facilitation Upper Extremity Pattern Exercises on Respiratory Functions, Body Image, Self-Esteem and Psychological State
Brief Title: Upper Extremity Pattern Exercises and Respiratory Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ozden Gokcek, Principal Investigator, Ege University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 08/2023
Record Dates: First submitted 2023-11-10; First posted 2023-11-18 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Healthy Individuals
Keywords: Reathing exercises; Body Image; Depression; Proprioceptive Neuromuscular Facilitation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: It includes a single-group exercise application with volunteer healthy university students.
Masking Description: The researcher who performed the evaluation did not participate in the exercise sessions applied in the study. He/she does not have information about the application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Group (Experimental): Proprioceptive neuromuscular facilitation upper extremity pattern exercises will be actively applied to 20 individuals in groups of 5 in a standing position for 30 minutes in each session 3 days a week for 4 weeks.
  Interventions: Other: Proprioceptive Neuromuscular Facilitation Upper Extremity Pattern

INTERVENTIONS:
Other: Proprioceptive Neuromuscular Facilitation Upper Extremity Pattern — Proprioceptive neuromuscular facilitation upper extremity pattern exercises will be actively applied to 20 individuals in groups of 5 in a standing position for 30 minutes in each session 3 days a week for 4 weeks.
  PNF upper extremity patterns to be applied to the participants:
  1. Bilateral symmetrical flexion-adduction-external rotation.
  2. Bilateral symmetrical flexion-abduction-external rotation.
  3. Bilateral asymmetric right: flexion-abduction-external rotation, left: flexion-adduction-external rotation.
  4. Bilateral reciprocal (same diagonal) right: extension-adduction-internal rotation, left: flexion-abduction-external rotation.
  5. Bilateral reciprocal (same diagonal) right: flexion-adduction-external rotation, left: extension-abduction-internal rotation.
  6. Bilateral reciprocal (opposite diagonal) right: extension-adduction-internal rotation, left: flexion, adduction, external rotation.

SUMMARY:
The study will be carried out with healthy students between the ages of 18-25 years who are studying at Ege University Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation and who voluntarily agree to participate in the study. Informed consent form will be signed before the evaluation of the individuals. The study will be carried out as a single group with the inclusion of a total of 20 individuals. The students who volunteered to participate in the study will actively apply the selected PNF upper extremity patterns for 4 weeks and will be evaluated twice, before and after the application. Demographic information of the individuals; age, height, weight, gender, background, surname, smoking habit, alcohol habit, education level (class), sports habit, COVID-19 disease status and when it occurred will be recorded. Cosmed pulmonary function test device will be used to evaluate the respiratory function of the individuals, Oncomed brand electronic body weight and height measurement device will be used to calculate the body mass index. Body Image Perception Scale will be used for body image perception, Beck Depression Inventory will be used to evaluate psychological status, and Rosenberg Self-Esteem Scale will be used to evaluate sense of self.

ELIGIBILITY:
Inclusion Criteria:

* Not diagnosed with any chronic disease
* No neurological problems
* Has not had COVID-19 for at least 6 months

Exclusion Criteria:

* Diagnosed with respiratory system diseases
* Regular medication use
* Suspected pregnancy
* Individuals with rheumatic or neurological diseases

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Forced vital capacity (FVC) | At the beginning and at the end of 4 weeks of exercise.
  It will be evaluated with Cosmed pulmonary function test device. The test will be performed according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria. The patient will be asked to take a deep breath in a sitting position and then exhale rapidly through the spirometer. Nasal clamp will be used during exhalation.
Forced expiratory volume in the first second (FEV1) | At the beginning and at the end of 4 weeks of exercise.
  It will be evaluated with Cosmed pulmonary function test device. The test will be performed according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria. The patient will be asked to take a deep breath in a sitting position and then exhale rapidly through the spirometer. Nasal clamp will be used during exhalation.
Forced expiratory volume in the first second/Forced vital capacity (FEV1/FVC) | At the beginning and at the end of 4 weeks of exercise.
  It will be evaluated with Cosmed pulmonary function test device. The test will be performed according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria. The patient will be asked to take a deep breath in a sitting position and then exhale rapidly through the spirometer. Nasal clamp will be used during exhalation.
Forced expiratory flow between 25% and 75% of vital capacity (FEF25-75) | At the beginning and at the end of 4 weeks of exercise.
  It will be evaluated with Cosmed pulmonary function test device. The test will be performed according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria. The patient will be asked to take a deep breath in a sitting position and then exhale rapidly through the spirometer. Nasal clamp will be used during exhalation.
Body Image Perception Scale | At the beginning and at the end of 4 weeks of exercise.
  The scale provides information about body image. The scale assesses satisfaction with 40 different body parts and functions. The scale has a minimum score of 40 and a maximum score of 200. A higher overall score on the scale indicates a higher negative judgement, while a lower overall score suggests a more positive evaluation.

SECONDARY OUTCOMES:
Rosenberg Self-Esteem Scale | At the beginning and at the end of 4 weeks of exercise.
  The scale consists of 63 items. It is evaluated over 12 subscales and it is accepted that those who score 0-1 on the self-esteem subscale have high self-esteem, those who score 2-4 have medium self-esteem and those who score 5-6 have low self-esteem.
Beck Depression Inventory | At the beginning and at the end of 4 weeks of exercise.
  It is a scale developed to measure the behavioural findings of depression. As a result of the scoring, 0-9 points are interpreted as Minimal, 10-16 points as Mild, 17-29 points as Moderate, 30-63 points as Severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Karsıyaka, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and the data repository containing the participants' data can be requested from the principal investigator upon valid requests. The corresponding author can be reached via e-mail.
Supporting Information: Study Protocol, SAP
Time Frame: Accessible for two years from the end of the study.